CLINICAL TRIAL: NCT06814860
Title: Microenvironmental Trial of Classical Hodgkin Lymphoma in Adolescents
Acronym: LH2004ME
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LH2004ME; RC-2022-2773380 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-01-02; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; adolescent; microenvironment; immune-check points
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin fixed paraffin embedded (FFPE) samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background. Classical Hodgkin's lymphoma (cHL) in adolescents between 15 and 18 years shows a higher disease-related mortality and the overall prognosis is worse than both children and adults.

Objectives. To investigate the immune checkpoint inhibitors (ICPI) therapeutic targets and specific T-regulatory and cytotoxic T-cell subsets, in the subgroup of adolescent cHL patients and to investigate their prognostic power.

Methods: Retrieved formalin-fixed paraffin-embedded (FFPE) of adolescent patients diagnosed with cHL with available clinical and tested by immunohistochemistry the immune checkpoint molecules CTLA-4, LAG-3, PD-1 and PDL1 and the biological markers FOXP3 and CD8.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 to 18 years at diagnosis of Classical Hodgkin lymphoma.

Exclusion Criteria:

* Unavailability/insufficiency of histological material for diagnosis.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 12 to 18 years who were histologically diagnosed with Classical Hodgkin lymphoma between 01/01/1996 and 31/12/2020 will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Characterization of the tumour microenvironment | through study completion, an average of 3 months
  Identification of phenotypic markers with possible prognostic and/or therapeutic impact predictive of clinical outcomes in patients undergoing LHC in pediatric/adolescent age.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sabattini, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy